CLINICAL TRIAL: NCT03709745
Title: A Randomized Trial Comparing Treatment with Aflibercept and Ranibizuamab for Macular Edema After Branch Retinal Vein Occlusion
Brief Title: Eylea and Lucentis for Macular Edema in Branch Retinal Vein Occlusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Erik Eye Hospital (Other)
Responsible Party: Principal Investigator, Anders Kvanta, Principal investigator, St. Erik Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/2422-31
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Branch Retinal Vein Occlusion with Macular Edema
MeSH Terms: interventions — aflibercept; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aflibercept (Active Comparator): Aflibercept is given monthly (at least 3 times) until resolution of macular edema after which the patient is observed monthly. If there is recurrence of macula edema, the patient is given aflibercept according to a treat-and-extend regimen.
  Interventions: Drug: Aflibercept Injection [Eylea]
- Ranibizumab (Active Comparator): Ranibizumab is given monthly (at least 3 times) until resolution of macular edema after which the patient is observed monthly. If there is recurrence of macula edema, the patient is given ranibizumab according to a treat-and-extend regimen.
  Interventions: Drug: Ranibizumab Injection [Lucentis]

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — Intravitreal injection is given as described in the arm description
  Other Names: Eylea
  Arms: Aflibercept
Drug: Ranibizumab Injection [Lucentis] — Intravitreal injection is given as described in the arm description
  Other Names: Lucentis
  Arms: Ranibizumab

SUMMARY:
Comparing time to recurrence of macular edema after an initial loading dose of at least three monthly anti VEGF injections (aflibercept or ranibizumab) for macular edema in BRVO.

DETAILED DESCRIPTION:
One hundred and ten patients with macular edema (ME) secondary to BRVO are randomized (1:1) to treatment with intravitreal injections of aflibercept or ranibizumab. An initial loading dose of at least three monthly injections is given in the study eye until the ME is resolved. Then patients are observed at regular intervals, initially every four weeks until study completion. Total follow-up time is nine months from baseline to completion. If ME recurs, patients are treated according to a treat-and-extend algorithm.

At every visit, visual acuity (VA) is measured with an ETDRS chart at 4 m. The fundus is examined by indirect ophthalmoscopy and by optical coherence tomography (OCT). Macular ischemia is evaluated with OCT angiography (OCT-A), visual field status with computerised perimetry and retinal sensitivity with microperimetry. Choroidal thickness is evaluated with enhanced depth imaging (EDI) OCT. Vision related quality of life (QoL) with NEI VFQ25.

ELIGIBILITY:
Inclusion Criteria:

* BRVO naïve patients, disease duration 1-6 months, BCVA 23-73 ETDRS letters (20/40-20/320), macula edema with intraretinal cysts and CRT > 300 micrometers (Cirrus)

Exclusion Criteria:

* BRVO with neovascular component, intraocular surgery during the previous 3 months, earlier vitreoretinal surgery, vascular retinopathy of other cause, intraocular infection/inflammation, myocardial infarction och cerebrovascular stroke during the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Difference in time to recurrence of macular edema | 9 months
  Time, in weeks, from completion of loading dose to first recurrence of macular edema.

SECONDARY OUTCOMES:
Comparison of the number of patients without ME in each treatment arm at one month after the first injection | 1 month
  The number of patients without macular edema at one month after the 1st injection in each treatment arm are compared
Comparison of the number of injections needed in each treatment arm to resolve ME | 9 months
  The number of injections needed for macular edema to resolve in each treatment arm are compared
Correlation between choroidal thickness and recurrence of ME and with non response to the treatment drugs. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Kvanta, MD PhD, Principal Investigator — St. Erik Eye Hospital
Locations (1):
- St Eriks Eye Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No